CLINICAL TRIAL: NCT07114380
Title: Investigation of Cold Snare Polypectomy for Removing 10-20 mm 0-Ip Colorectal Polyp: One Feasibility and Safety Study
Brief Title: Investigation of Cold Snare Polypectomy for Removing 10-20 mm 0-Ip Colorectal Polyp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202505029RINA
Record Dates: First submitted 2025-07-20; First posted 2025-08-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: 10-20 mm Pedunculated Colorectal Polyp
Keywords: cold snare polypectomy; pedunculated polyp; efficacy; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cold snare polypectomy (Experimental): Participants in this single-arm study will undergo cold snare polypectomy (CSP) for removal of 10-20 mm pedunculated colorectal polyps identified during clinically indicated colonoscopy. CSP will be performed using standard cold snares without electrocautery. The procedure will be conducted by experienced endoscopists, and all peri-procedural care will follow routine clinical protocols. Outcomes will include complete resection rate, procedure time, and occurrence of adverse events such as immediate or delayed bleeding, perforation, and emergency visits.
  Interventions: Device: Cold snare polypectomy

INTERVENTIONS:
Device: Cold snare polypectomy — Unlike traditional hot snare polypectomy or endoscopic mucosal resection, which use electrocautery to resect larger or pedunculated polyps, cold snare polypectomy uses mechanical transection alone without cautery. The procedure is performed using a dedicated cold snare by experienced endoscopists.

SUMMARY:
This is a multicenter, single-arm feasibility study conducted across multiple hospitals in Taiwan. The goal of this trial is to evaluate whether cold snare polypectomy is a feasible and safe method for removing 10-20 mm pedunculated colorectal polyps.

The main questions it aims to answer are:

1. Can cold snare polypectomy achieve complete removal of 10-20 mm pedunculated polyps?
2. What are the rates and types of complications associated with this technique?

Participants will:

1. Undergo colonoscopy as clinically indicated
2. Have 10-20 mm pedunculated polyps removed using cold snare polypectomy if eligible
3. Be monitored for post-procedure outcomes, including pathology results and any complications

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm clinical trial designed to evaluate the feasibility and safety of cold snare polypectomy (CSP) for the removal of 10-20 mm pedunculated (0-Ip) colorectal polyps. While CSP is widely recommended for polyps <10 mm due to its favorable safety profile and comparable efficacy to hot snare polypectomy (HSP), its application for larger pedunculated polyps remains insufficiently studied, particularly given concerns regarding bleeding risk.

The study will enroll 120 adult participants undergoing colonoscopy at one of five hospitals in Taiwan. Participants found to have 10-20 mm 0-Ip polyps that are deemed amenable to CSP will undergo cold snare resection by experienced endoscopists. Standard pre- and post-procedure care will be followed. Polyp characteristics, resection outcomes, and complications (e.g., immediate or delayed bleeding, perforation, emergency visits) will be recorded.

Primary endpoints include technical success (complete removal as assessed by endoscopy and pathology) and safety (rate of adverse events such as bleeding or perforation). Clinical and procedural data will be collected prospectively, and statistical analysis will be conducted to identify predictors of CSP failure using univariate and multivariate models.

This study aims to fill a critical knowledge gap in the literature regarding the appropriateness of CSP for larger pedunculated lesions and inform future guideline recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Undergoing colonoscopy for any clinical indication
* Found to have a 10-20 mm pedunculated colorectal polyp suitable for cold snare polypectomy

Exclusion Criteria:

* Age < 20 years
* Medical contraindications to colonoscopy or polypectomy (e.g., recent myocardial infarction, stroke, severe unstable cardiovascular disease, acute peritonitis, fulminant colitis, perforation, or toxic megacolon)
* Inadequate bowel preparation preventing complete colonoscopy or safe polypectomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Cold snare polypectomy successful resection rate | From the start of the colonoscopy to completion of the procedure, typically within 1 hour)
  The investigators will record whether each polyp is removed by cold snare polypectomy with or without resistance. These will be considered successful resection cases. Polyps that cannot be removed by cold snare polypectomy and require switching to hot snare polypectomy will be considered failed resection cases.

SECONDARY OUTCOMES:
Number of Polyps with Immediate Bleeding After Cold Snare Polypectomy | From the start of the colonoscopy to completion of the procedure, typically within 1 hour.
  Definition: Immediate bleeding would be assessed and graded during the procedure. The severity grades were listed as followed,
  1. Grade 1: Spontaneous hemostasis within 1 minute
  2. Grade 2: Continuous but decreased oozing over 1 minute
  3. Grade 3: Continuous oozing over 1 minute
  4. Grade 4: Active spurting
  Unit of Measure: Number of polyps with immediate bleeding, stratified by grade
Number of Participants with Delayed Bleeding After Cold Snare Polypectomy | From completion of colonoscopy until the date of first documented event, assessed up to 14 days post-procedure.
  Definition: Any bleeding episode occurring after the patient has left the endoscopy unit and within 14 days post-polypectomy, classified as:
  Mild: Bleeding stops spontaneously without medical intervention
  Severe: Hemoglobin drop >2 g/dL from baseline, need for blood transfusion, or requirement of endoscopic, angiographic, or surgical hemostasis
  Unit of Measure: Number of participants with delayed bleeding
Number of Participants with Perforation | From start of colonoscopy until the date of first documented event, assessed up to 14 days post-procedure.
  Definition: Any full-thickness defect of the colonic wall identified during or after the procedure.
  Unit of Measure: Number of participants with perforation
Number of Participants with Post-Polypectomy Emergency Department Visits | From start of colonoscopy until the date of first documented event, assessed up to 14 days post-procedure.
  Definition: Any unplanned emergency department visit related to post-polypectomy complications.
  Unit of Measure: Number of participants with emergency department visits
Polypectomy time | From the start of the colonoscopy to completion of the procedure, typically within 1 hour.
  Description: Time from when the snaring instrument first appears on the colonoscopy screen to when colonoscope withdrawal resumes after polypectomy.
  Unit of Measure: Seconds
Withdrawal Time | From the start of the colonoscopy to completion of the procedure, typically within 1 hour.
  Description: Total time taken to withdraw the colonoscope from cecum to anus
  Unit of Measure: Minutes
Number of Polyps with En Bloc Resection | From the start of the colonoscopy to completion of the procedure, typically within 1 hour.
  Description: Whether the polyp was removed in a single piece (en bloc).
  Unit of Measure: Number of polyps with en bloc resection
Number of Polyps with Complete Histologic Resection | From end of colonoscopy exam to pathology report, usually within 2 weeks.
  Description: Whether pathology confirms tumor-free margins in the resected specimen.
  Unit of Measure: Number of polyps with complete histologic resection
Number of Polyps Requiring Prophylactic Hemoclipping | From the start of the colonoscopy to completion of the procedure, typically within 1 hour.
  Description: Whether hemoclips were applied prophylactically after cold snare polypectomy.
  Unit of Measure: Number of polyps requiring prophylactic hemoclipping
Number of Polyps Requiring Submucosal Injection | From the start of the colonoscopy to completion of the procedure, typically within 1 hour.
  Description: Whether submucosal injection was required before or during cold snare polypectomy.
  Unit of Measure: Number of polyps requiring submucosal injection
Number of Polyps Successfully Retrieved | From the start of the colonoscopy to completion of the procedure, typically within 1 hour.
  Description: The number of resected polyps that are successfully retrieved and submitted for histologic evaluation.
  Unit of Measure: Number of polyps successfully retrieved

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chun Chang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - National Taiwan University Hospital, Jinshan Branch, New Taipei City
  - National Taiwan University Cancer Center, Taipei
  - National Taiwan University Hospital, Bei-Hu Branch, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tseng CH, Chang LC, Wu JL, Chang CY, Chen CY, Chen PJ, Shun CT, Hsu WF, Chen YN, Chen CC, Huang TY, Tu CH, Chen MJ, Chou CK, Lee CT, Chen PY, Lin JT, Wu MS, Chiu HM. Bleeding Risk of Cold Versus Hot Snare Polypectomy for Pedunculated Colorectal Polyps Measuring 10 mm or Less: Subgroup Analysis of a Large Randomized Controlled Trial. Am J Gastroenterol. 2024 Nov 1;119(11):2233-2240. doi: 10.14309/ajg.0000000000002847. Epub 2024 May 9. PMID 38775310
- [Background] Ferlitsch M, Hassan C, Bisschops R, Bhandari P, Dinis-Ribeiro M, Risio M, Paspatis GA, Moss A, Libanio D, Lorenzo-Zuniga V, Voiosu AM, Rutter MD, Pellise M, Moons LMG, Probst A, Awadie H, Amato A, Takeuchi Y, Repici A, Rahmi G, Koecklin HU, Albeniz E, Rockenbauer LM, Waldmann E, Messmann H, Triantafyllou K, Jover R, Gralnek IM, Dekker E, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2024. Endoscopy. 2024 Jul;56(7):516-545. doi: 10.1055/a-2304-3219. Epub 2024 Apr 26. PMID 38670139
- [Background] Kaltenbach T, Anderson JC, Burke CA, Dominitz JA, Gupta S, Lieberman D, Robertson DJ, Shaukat A, Syngal S, Rex DK. Endoscopic Removal of Colorectal Lesions-Recommendations by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1095-1129. doi: 10.1053/j.gastro.2019.12.018. Epub 2020 Feb 11. No abstract available. PMID 32122632
- [Background] Copland AP, Kahi CJ, Ko CW, Ginsberg GG. AGA Clinical Practice Update on Appropriate and Tailored Polypectomy: Expert Review. Clin Gastroenterol Hepatol. 2024 Mar;22(3):470-479.e5. doi: 10.1016/j.cgh.2023.10.012. Epub 2023 Nov 28. PMID 38032585
- [Background] Qu J, Jian H, Li L, Zhang Y, Feng B, Li Z, Zuo X. Effectiveness and safety of cold versus hot snare polypectomy: A meta-analysis. J Gastroenterol Hepatol. 2019 Jan;34(1):49-58. doi: 10.1111/jgh.14464. Epub 2018 Sep 26. PMID 30176072
- [Background] Chang LC, Chang CY, Chen CY, Tseng CH, Chen PJ, Shun CT, Hsu WF, Chen YN, Chen CC, Huang TY, Tu CH, Chen MJ, Chou CK, Lee CT, Chen PY, Wu MS, Chiu HM. Cold Versus Hot Snare Polypectomy for Small Colorectal Polyps : A Pragmatic Randomized Controlled Trial. Ann Intern Med. 2023 Mar;176(3):311-319. doi: 10.7326/M22-2189. Epub 2023 Feb 21. PMID 36802753